CLINICAL TRIAL: NCT03362229
Title: Medial Malleolus: Operative or Non-operative - A Prospective Randomized Controlled Trial of Operative Versus Non-operative Management of Associated Medial Malleolus Fractures in Unstable Fracture Dislocations of the Ankle Joint'
Brief Title: Medial Malleolus: Operative Or Non-operative
Acronym: MOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Tom Carter, Principle Investigagor, Royal Infirmary of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/0262
Record Dates: First submitted 2017-11-09; First posted 2017-12-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Ankle Fracture - Medial Malleolus
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with 50:50 randomisation into one of 2 groups. Randomisation will also be stratified be age of patient (>= 65 and <65 years).
Masking Description: There is no blinding possible in this trial as the presence or absence of medial sided surgery is obvious to both the surgeon and the patient due to the presence or absence of a skin incision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FIXATION (Active Comparator): Medial malleolus fixation, with the method of fixation left to the surgeons discretion.
  Interventions: Procedure: Fixation
- NON-FIXATION (Active Comparator): A well reduced medial malleolus fracture is then left without fixation ie, non-operative management.
  Interventions: Procedure: Non-fixation

INTERVENTIONS:
Procedure: Fixation — A well reduced medial malleolus fracture will undergo internal fixation, guided by the surgeon's skill and expertise
  Arms: FIXATION
Procedure: Non-fixation — A well reduced medial malleolus fracture will be left without fixation
  Arms: NON-FIXATION

SUMMARY:
Medial malleolus: Operative Or Non-operative (MOON study) Ankle fractures are a common Orthopaedic trauma presentation, accounting for approximately 10% of the workload. There has been debate regarding the significance of the contribution of the medial malleolus to ankle stability. Some deem the lateral malleolus as the key stabiliser. With this anatomically aligned the ankle joint should be stable. Operating on the medial malleolus fracture often requires a second generous skin incision, soft tissue stripping and insertion of metalwork. This carries with it the risk of wound complications, infection and increased operation time. High risk patients including the elderly, diabetics and those with significant swelling following injury are particularly vulnerable. The study will include adult patients (≥16 years) with capacity to consent and complete post-operative questionnaires, presenting to a single Orthopaedic trauma unit. Participants will be randomised to fixation or non-fixation of associated medial malleolus fractures at the same time as fixation of the lateral malleolar fracture to assess if this impacts on validated patient outcomes, failure, operative time and complications over a one-year follow-up. Only one trial has been published, showing no significant difference between failure rates or outcomes, but reduced operative time.

Participants will be enrolled into the trial following informed consent. The final decision on whether a participant is eligible can only be made during surgery when the medial malleolus fracture has reduced with no more than 2mm displacement. If this is confirmed the participant will be randomised to receive either fixation or non-fixation of the medial malleolus. Randomisation therefore occurs at the time of surgery. Participants will be reviewed at set post-operative checkpoints, with X-rays and patient reported outcome scores. Trial data will hopefully enable surgeons to make better informed decisions when managing patients with ankle fracture dislocations.

DETAILED DESCRIPTION:
This trial will include adult patients (16 years) presenting to the single centre; Edinburgh Orthopaedic Trauma Unit, Royal Infirmary of Edinburgh, with an isolated unstable fracture of the ankle joint requiring operative intervention. Both NHS research ethics committee (REC) approval and NHS R&D Management approval have been granted.

All patients will be treated in the Emergency Department (ED) with closed reduction and casting under procedural sedation and then referred to Orthopaedics via the on-call service. Patients will be considered for the trial if the following criteria are met:

1. Aged 16 years or older.
2. An unstable fracture dislocation of the ankle joint, defined as a bimalleolar or trimalleolar fracture pattern with or without any of the following:

   * Radiographic evidence of talar shift
   * Posterior malleolar fracture of >25% articular involvement or >2mm step-off
   * Syndesmosis injury

Patients who consent to participate in the trial will be enrolled into the trial pre-operatively, but the result of their randomisation will not be revealed until after fibular fixation and assessment of medial malleolus reduction intra-operatively. Patients will only be eligible to continue in the trial if the medial malleolus reduces to acceptable limits without open reduction (≤2mm of displacement as seen on a radiographic antero-posterior view). If the medial malleolus fracture does not reduce within this 2mm limit, the patient will require formal open reduction and internal fixation and consequently not suitable to continue in the trial. The inclusion and exclusion criteria for this trial are displayed below.

Vulnerable populations, including patients unable to give consent and complete post-operative questionnaires, will not be recruited. A participant information sheet will be provided for them to read before agreeing to take part. The study protocol will then be reviewed in detail and a member of the research team member will complete the informed consent process. With the permission of the patient, a letter will be sent to their General Practitioner informing them of their involvement in the trial and patients will be given a copy of their consent form. Patients may take as long as they like to consider participation, provided that they still meet all the eligibility criteria documented above. Patients who require additional time to make a decision will be contacted the following day by a further face-to-face inpatient discussion. They will also be given the contact details of an Orthopaedic specialist, independent of the trial to allow them access to further information if they require. Upon agreeing to take part, participants will be randomised into one of two treatment groups intra-operatively by closed opaque envelope: operative or non-operative management of the medial malleolus fracture. Randomisation will be stratified according to age to allow an even distribution of both young (<65 years) and older (65+ years) patients between the operative groups. The result of their randomisation will only be revealed if the fracture reduces spontaneously following lateral malleolus fixation with ≤2mm of residual displacement. On enrolment, a data collection form will be started with demographic and injury-related information collected. Regardless of the treatment allocation, the patients will be followed up at the following post-operative stages: 2 weeks, 6 weeks, 3 months, 6 months and one year. This will be either in person in the outpatient clinic or via postal questionnaire. At each visit physical examination, treatment, complications and re-operation (e.g. hardware removal) for each patient will be recorded. Participants will be asked to complete their outcome scores independently, as they would with the postal questionnaires. The presence or absence of a medial sided incision and obvious differences with respect to metalwork on radiographs means neither the patient nor the investigator can be blinded to the treatment group. The investigators will also follow up patients' records to assess whether they underwent any subsequent surgery on the affected ankle during the study period. This would include debridement/irrigation for infection and/or removal of metalwork for a variety of reasons.

Interventions - Patients randomised to operative management of the associated medial malleolus fracture will be treated routinely with standard medial malleolus fixation techniques. The most common being the use of 2x 3.5mm partially threaded cancellous screws (35mm - 45mm length) inserted at 90 degrees to the fracture line, following satisfactory open reduction. Other techniques, used far less frequently include the use of a tension band wire construct and Kirschner wires. The technique employed will be at the discretion of the treating surgeon and aims to reproduce the decisions that are made in day-to-day trauma care. Those participants who are not suitable for randomisation intra-operatively as the medial malleolus does not reduce within acceptable limits will be excluded from the trial. The result of their randomisation will not be revealed and their envelope will be return to the study office and allocated in order to the next eligible patient. This will limit disruption to the randomisation sequence. The subsequent care of that patient will then be at the discretion of their treating consultant.

Post-operative immobilisation and weight bearing restrictions will be at the discretion of the treating surgeon, which again reflects everyday practice when managing this common orthopaedic injury. However, the default immobilisation will be in a removable supportive orthosis (walking boot) and patients will be allowed to fully weight bear unless there is a clinical indication, as highlighted above. Post-operative physiotherapy will be arranged at the discretion of the treating surgeon, as occurs in routine clinical practice.

Power analysis - Prior to the study a power analysis determined the number of patients required in each arm of the trial. The primary outcome measure will be the OMAS at one year. To show a clinically meaningful difference in means OMAS at one year between the groups of 10 points, assuming a common standard deviation of 20 points, 80% power and 5% level of significance the study would require 64 participants per groups (i.e. a total of 128). However, to account for potential dropouts through the duration of the study this number will increase by 20% to 77 per group (i.e. a total of 154).

Statistical analysis for the trial will be performed by an independent statistician employed through the local University statistics department/Edinburgh Clinical Research Facility. Primary and secondary outcome measures are displayed in the relevant section below.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 years
2. Able to consent to treatment
3. Unstable fracture dislocation of the ankle joint requiring operative intervention as defined in section 3.1
4. Closed injury
5. Weber B & Weber C fractures
6. Surgery date within two weeks of date of fracture

Exclusion Criteria:

1. Patients unable to comply with post-operative data gathering including completing questionnaires in English language
2. Additional lower limb injury, which may impact on patient rehabilitation
3. Open fracture
4. Confirmed severe associated neurovascular injuries
5. Distal tibial intra-articular fractures/ pilon type injuries
6. Supination-adduction type 2 (SAD-2) fracture configurations with a medial malleolus vertical shear fracture
7. Patients medically unfit for surgery
8. Patients declining operative management
9. Non-residents, unable to return to the unit for follow-up for a period of 1-year
10. Current engagement in a pharmaceutical/drug trial
11. Where the treating surgeon does not feel that inclusion in the trial is in the patients' best interest either due to the fracture pattern or patient factors

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — We hypothesise we will recruit slightly more females than males as this is our experience in our local unit with routine practice.
Enrollment: 154 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Olerud & Molander Ankle Score (OMAS) over a one-year post-operative period | 6 week, 3 months, 6 months and one year.
  The OMAS is a functional rating scale developed in 1984, which has been used extensively as a research tool in foot and ankle surgery. It includes nine parameters: pain, stiffness, swelling, stair climbing, running, jumping, squatting, supports and work/activities of daily living. The sub-score parameters are summated to generate a final score from 0 - 100, with '100' representing an excellent functional outcome and '0' being the worse possible outcome.

SECONDARY OUTCOMES:
Change in Euroqol-5D over a one-year post-operative period | 6 week, 3 months, 6 months and one year.
  A standardised instrument for use as a measure of health outcome. A score of '+1.0' represents an excellent state of general health and a score of '-1.0' represents a very poor state of general health.
Change in Manchester-Oxford Foot Questionnaire (MOXFQ) over a one-year post-operative period | 6 week, 3 months, 6 months and one year.
  A validated and reliable PROM for surgery of the foot and ankle, it consists of 16-items from three domains: walking/standing (7 items), pain (5 items) and social interaction (4 items). Each item is scored on a 5-point Likert scale ranging from no limitation to maximum limitation (0,1,2,3,4). The sub-scales are summated to generate a raw score out of 64 is then converted to a 0 - 100 metric score, with '100' being awarded for the most severe limitation and a score of '0' for no limitation whatsoever.
Tourniquet time | Immediately post-operatively
  Length of time tourniquet inflated for during surgery
Change in Visual analogue pain scale (VAS) over a one-year post-operative period | 6 week, 3 months, 6 months and one year.
  Assessment of pain with '100' being no pain and '0' being extreme pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Edinburgh Orthopaedic Trauma Unit, Edinburgh Royal Infirmary, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carter TH, Oliver WM, Bell KR, Graham C, Duckworth AD, White TO. Operative vs Nonoperative Management of Unstable Medial Malleolus Fractures: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2351308. doi: 10.1001/jamanetworkopen.2023.51308. PMID 38236603
- [Derived] Carter TH, Oliver WM, Graham C, Duckworth AD, White TO. Medial malleolus: Operative Or Non-operative (MOON) trial protocol - a prospective randomised controlled trial of operative versus non-operative management of associated medial malleolus fractures in unstable fractures of the ankle. Trials. 2019 Sep 12;20(1):565. doi: 10.1186/s13063-019-3642-7. PMID 31514744